CLINICAL TRIAL: NCT00210496
Title: Efficacy of AXERT (Almotriptan Malate) in the Acute Treatment of Migraine: A Pilot Study of the Potential Impact of Preventive Therapy With TOPAMAX (Topiramate)
Brief Title: Potential Impact (Benefit) of Preventative Treatment With Topamax on the Effectiveness of Axert in the Acute Treatment of Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Ortho LLC (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002875
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Migraine; Classic Migraine; Common Migraine
Keywords: Migraine headache; Topiramate, Almotriptan malate
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura | interventions — Topiramate; almotriptan

INTERVENTIONS:
Drug: topiramate; almotriptan malate

SUMMARY:
The purpose of this study is to evaluate the impact of topiramate (migraine prevention medicine) on the effectiveness of almotriptan malate (acute migraine medicine) when treating acute migraine headaches.

DETAILED DESCRIPTION:
Migraine afflicts greater than 28 million adults in the United States. Acute treatments, such as almotriptan malate, target the symptoms of a migraine attack. Preventive treatments, such as topiramate, primarily target the generation of attacks and may decrease use of acute treatments. Preventive treatments, by a process of neurostabilization, may result in an additive effect on almotriptan malate to improve acute treatment intervention response during a migraine attack. This is a randomized, double blind, parallel group multicenter study that will enroll patients 18-65 years old with a history of 3-12 migraine headaches each month for the past 3 months. The total study duration will be approximately 32 weeks. The study is divided into 4 phases as follows: A Screening Phase that lasts one month; An Open Label Phase where all patients will be treated with topiramate gradually dosed to 100mg a day lasting 6 weeks; A Double Blind Phase lasting 19 weeks at which time patients will be randomized to stay on topiramate 100mg per day or switch to placebo topiramate (50:50 chance) and a Taper/Exit Phase lasting 2 weeks. Almotriptan malate will be used for all migraine headaches during the study as needed. The study hypothesis is that the combination of almotriptan malate and topiramate will have a better clinical response than the combination of almotriptan malate and placebo topiramate. Migraine pain information will be collected from each patient with the use of a Personal Digital Assistant (PDA or Palm Pilot) throughout the study for each migraine attack. Commercial Topiramate will be gradually increased to 100mg/day in approximately 4-6 weeks. You will then be randomized to either Topiramate or Placebo, dosed at 100mg a day, for the remainder of the study (18 weeks). AXERT 12.5mg may be taken to treat migraine headaches during the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of migraine headaches for at least 6 months
* Experience 3-12 migraines per month
* Able to take oral medication
* Able to complete the electronic diary (Personal Digital Assistant-PDA).

Exclusion Criteria:

* You will not be able to participate in the study if you previously discontinued Topiramate or Almotriptan because it did not make you feel better or it made you feel different
* Have 15 or more headache days a month
* Experience migraine aura without a headache
* Already on a migraine preventative medicine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2005-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness parameter will be the proportion of subjects in each treatment group who achieve a Sustained Pain Free (SPF) response during the first qualifying headache of the Assessment Period.

SECONDARY OUTCOMES:
For first headache of the Assessment Period, Pain relief at 2 hours; Pain free at 2 hours; Maximum intensity of headache pain; Headache duration; Rescue medication use; Maximum intensity of migraine associated symptoms (photophobia, phonophobia, nausea).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Ortho LLC Clinical Trial, Study Director — Janssen-Ortho LLC

REFERENCES:
- See also: Acute Treatment of Migraine Impact of Preventive Therapy w/TPM — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=291&filename=CR002875_CSR.pdf